CLINICAL TRIAL: NCT05479994
Title: A Single-Arm, Open-Label, Multicenter Phase 2 Study to Evaluate the Efficacy and Safety of BCL2 Inhibitor BGB-11417 in Adult Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: Study of BGB-11417 in Participants With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-202; CTR20222085 (Other: ChinaDrugTrials)
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Leukemia; Lymphoma; Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Small Lymphocytic Lymphoma; Relapsed Chronic Lymphocytic Leukemia
Keywords: Refractory Chronic Lymphocytic Leukemia; Leukemia; Lymphoma; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Participants will receive BGB-11417 orally until disease progression, intolerable toxicity, or other scenarios specified in the protocol
  Interventions: Drug: BGB-11417

INTERVENTIONS:
Drug: BGB-11417 — Administered orally
  Other Names: sonrotoclax

SUMMARY:
The purpose of this study is to evaluate the efficacy of BGB-11417 in participants with relapsed/refractory (R/R) chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL)

ELIGIBILITY:
Key Inclusion Criteria

1. Participants with a histologically confirmed diagnosis of CLL/SLL based on the International Workshop on CLL (iwCLL) criteria:

   1. Treatment intolerance or failure during or after treatment with chemoimmunotherapy (CIT) and BTK inhibitors (BTKi) or
   2. Treatment intolerance or failure during or after treatment with BTKi for CIT-ineligible participants as assessed by the investigator.
2. Participants who require treatment based on the iwCLL 2018 criteria
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 2
4. Life expectancy of > 6 month

Key Exclusion Criteria

1. Prior malignancy within the past 2 years, except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or low risk (Gleason score ≤ 6) localized prostate cancer
2. Underlying medical conditions that, in the investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of safety or efficacy results
3. A known history of or currently suspected Richter's syndrome
4. Prior autologous stem cell transplant (unless ≥ 3 months after transplant) or prior chimeric cell therapy (unless ≥ 6 months after cell infusion)
5. Prior allogeneic stem cell transplant

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) as assessed by the Independent Review Committee (IRC) | Up to 2 Years
  Defined as the proportion of participants who achieved a complete response (CR), complete remission with incomplete marrow recovery (CRi), nodular partial response (nPR), or partial response (PR) per the 2018 iwCLL guidelines for participants with chronic lymphocytic leukemia (CLL) or Defined as the proportion of participants who achieved PR or better per the Lugano Classification for partiticpants with small lymphocytic lymphoma (SLL)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) as assessed by the investigator | Up to 2 Years
  Defined as the proportion of participants who achieved a complete response (CR), complete remission with incomplete marrow recovery (CRi), nodular partial response (nPR), or partial response (PR) per the 2018 iwCLL guidelines for participants with chronic lymphocytic leukemia (CLL) or Defined as the proportion of participants who achieved PR or better per the Lugano Classification for participants with small lymphocytic lymphoma (SLL)
Duration of response (DoR) as determined by the IRC and the investigator | Up to 5 Years
  DoR is defined as the time from first determination of response until first documentation of progression or death, whichever occurs first
Progression Free Survival (PFS) as determined by the IRC and the investigator | Up to 5 Years
  PFS is defined as the time from the date of the first study dose until the date of first documented disease progression or death due to any cause, whichever occurs first.
Time to Response (TTR) as assessed by investigator and IRC | Up to 2 Years
  TTR is defined as the time from treatment initiation to the first documented response.
Overall Survival (OS) | Up to 5 Years
  defined as time from the start of treatment to the date of death due to any cause
Participants Reported Outcome as measured by EQ-5D-5L questionnaires | Up to 5 Years
  The EQ-5D-5L descriptive system assesses health in five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT, ANXIETY / DEPRESSION), each of which has five levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to).
Participant Reported Outcomes as measured by NFLymSI-18 | Up to 5 Years
  The National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Lymphoma Cancer Symptom Index-18 (NFLymSI-18) questionnaire contains 18 items, each of which utilizes a Likert scale with 5 possible responses ranging from 0 'Not at all' to 4 'Very much' and is divided into a total score.
Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 5 Years
  with adverse events leading to discontinuation, and AEs graded according NCI-CTCAE Version 5 and the Grading Scale for Hematologic Toxicity in CLL Studies
Number of participants with clinically significant changes from baseline in vital signs | Up to 5 Years
  Vital signs include systolic and diastolic blood pressure, heart rate, and body temperature
Number of participants with clinically significant changes from baseline in clinical laboratory values | Up to 5 Years
  Laboratory values include hematology, clinical chemistry, coagulation, and urinalysis
Number of Participants With Clinically Significant Physical Examination Findings | Up to 5 Years
  A full physical examination includes head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal and musculoskeletal systems

CONTACTS AND LOCATIONS:
Locations (50):
- China (50):
  - Anhui Provincial Cancer Hospital Aka West Branch of Anhui Province Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University(Tongzhou), Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Quanzhou First Affliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - The Second Affiliated Hospital of Fujian Medical University Donghai Campus, Quanzhou, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Yuebei Peoples Hospital, Shaoguan, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Red Cross Hospital of Yulin City, Yulin, Guangxi
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hainan Cancer Hospital, Haikou, Hainan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University South Campus, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Northern Jiangsu Peoples Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Tonghua Center Hospital, Tonghua, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shaanxi Provincial Peoples Hospital, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Jining No Peoples Hospital West Branch, Jining, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The Third Peoples Hospital of Datong, Datong, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Dazhou Central Hospital, Dazhou, Sichuan
  - Peoples Hospital of Deyang City, Deyang, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - The First Peoples Hospital of Kashgar, Kashgar, Xinjiang
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/